CLINICAL TRIAL: NCT01537744
Title: Phase I Trial of Oral 5-azacitidine With Romidepsin in Advanced Solid Tumors, With an Expansion Cohort in Virally Mediated Cancers and Liposarcoma
Brief Title: A Trial of Oral 5-azacitidine in Combination With Romidepsin in Advanced Solid Tumors, With an Expansion Cohort in Virally Mediated Cancers and Liposarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J11102; NA_00052054 (Other: JHMIRB)
Record Dates: First submitted 2012-02-08; First posted 2012-02-23 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Solid Tumors; Virally Mediated Cancers and Liposarcoma
Keywords: expansion cohort
MeSH Terms: conditions — Liposarcoma | interventions — romidepsin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oral 5-azacitidine + romidepsin (Experimental): oral 5-azacitidine in combination with romidepsin
  Interventions: Drug: oral 5-azacitidine in combination with romidepsin

INTERVENTIONS:
Drug: oral 5-azacitidine in combination with romidepsin — DOSING REGIMEN(S):
  Table 1: Dose Escalation Schedule Dose Level Dose and Schedule a, c 5-Azacitidine (PO) Romidepsin (IV)
  Level -1b 100mg daily days 1-14 8mg/m2 days 8 and 15
  Level 1 200mg daily days 1-14 8mg/m2 days 8 and 15
  Level 2 300mg daily days 1-14 8mg/m2 days 8 and 15
  Level 3 300mg daily days 1-21 8mg/m2 days 8 and 15
  Level 4d MTD 8mg/m2 days 8, 15, and 22
  1. Each cycle will last 28 days.
  2. Subjects will be enrolled in Level -1 if the MTD is reached in the subjects enrolled in Level 1.
  3. On days when both agents are administered, oral 5-azacitidine should be administered at the start of the romidepsin infusion.
  4. Level 4 is optional and decisions whether to initiate this level will be based on discussions between the study investigator and Celgene.
  Other Names: 5-azacytidine; Vidaza; Istodax

SUMMARY:
The purpose of this study is to determine whether 5-azacitidine in combination with romidepsin cancer are effective in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is a two part, single-institution, open-label, Phase I dose-escalation study of oral 5-azacitidine in combination with intravenous (IV) romidepsin. Part 1 of the study is a traditional 3 + 3 dose escalation study designed to evaluate the maximum tolerated dose (MTD), dose limiting toxicities (DLTs), safety, pharmacokinetic (PK) profiles, and pharmacodynamic profiles of increasing doses of orally administered 5-azacitidine in combination with a constant dose of IV romidepsin. Part 2 is an expansion cohort study for the preliminary evaluation of efficacy in the treatment of virally mediated cancers and liposarcoma once the MTD has been determined. PK and PD data will also be collected for these subjects.

* Plasma samples will be obtained, prior and during treatment, to assess the methylation status of free tumor DNA circulating in the blood
* Archival tissue will be obtained on all participants for future correlative studies, such as baseline gene expression, methylation patterns.
* Participants with accessible, biopsiable tumors will also undergo pre-treatment and post-treatment (~cycle 2D1) biopsies for correlative studies in the expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign informed consent form (ICF).
* Age ≥ 18 years at time of signing ICF.
* Adhere to study visit schedule and other protocol requirements.
* Histologically or cytologically confirmed metastatic or unresectable solid tumor (phase I dose escalation), OR HPV+ nasopharyngeal cancer, HPV+ cervical cancer or liposarcoma (for expansion cohort).
* Failed at least one previous chemotherapy regimen for metastatic disease if standard therapies exist.
* Measurable disease per RECIST 1.1
* Life expectancy ≥ 12 weeks
* No previous cancer therapy ≥ 4 weeks.
* ECOG performance status ≤ 1
* Laboratory test results:

  * Absolute neutrophil count ≥ 1500/mm³
  * Platelet ≥ 100,000/mm³
  * Serum creatinine levels < 1.5 X ULN OR creatinine clearance >60 mL/min/1.73 m2 for subjects with creatinine levels > institutional normal
  * Serum bilirubin ≤ 1.5 times the upper limit of the normal range for the laboratory (ULN).
  * AST (SGOT) and ALT (SGPT) ≤ to 2.5 x ULN
* Disease free of prior malignancies ≥ 5 years (except currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast).
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with 5-azacitidine. All men/women of childbearing potential must use acceptable methods of birth control throughout the study.

Exclusion Criteria:

* Serious medical conditions, laboratory abnormality, or psychiatric illness that would prevent the subject from signing ICF.
* Pregnant or breastfeeding women. (Lactating women must agree not to breast feed while taking 5-azacitidine).
* Conditions, including laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret study data.
* Chemotherapy, radiotherapy, or experimental drug or therapy ≤ 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to enrollment or adverse events < grade 1 due to agents administered >4 weeks earlier except for stable grade 2 neuropathy.
* No other concomitant investigational agents.
* Known or suspected hypersensitivity to 5-azacitidine, romidepsin, mannitol or other agents used in this study.
* Uncontrolled brain metastases.
* Known positive for HIV, infectious hepatitis, type B or C.
* Uncontrolled intercurrent illness
* Known GI disorders precluding oral administration of 5-azacitidine.
* Known cardiac abnormalities such as:

  * Congenital long QT syndrome
  * QTc interval ≥ 500 milliseconds;
  * Myocardial infarction ≤6 months of C1D1. Subjects with a history of myocardial infarction between 6-12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate;
  * Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min);
  * Symptomatic coronary artery disease (CAD), e.g., angina. In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * Screening ECG showing evidence of cardiac ischemia (ST depression, depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI;
  * Known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
  * Hypertrophic cardiomegaly or restrictive cardiomyopathy;
  * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria; or
  * Cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
* Patients taking drugs leading to significant QT prolongation
* Concomitant use of CYP3A4 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From first dose of study treatment to end of study visit, approximately 1.5 years
  Incidence of adverse events, serious adverse events, and dose-limiting adverse events graded according to NCI CTCAE version 4
Maximum Tolerated Dose (MTD) | First cycle
  MTD defined as the highest dose level at which < 2 out of 6 patients experienced a DLT.
Clinical responses associated with oral 5-azacitidine and romidepsin | Measured every two cycles during study treatment, expected duration ≤1.5 years
  Clinical responses associated with oral 5-azacitidine and romidepsin treatment in subjects with advanced solid malignancies according to RECIST criteria [Time Frame: measured every two cycles during study treatment, expected duration ≤1.5 years

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | On Day 1 and 8 of Cycle 1
  Peak plasma concentration (Cmax), area under the concentration versus time curve (AUC) from time 0-infinity, elimination half-life (t1/2), clearance, and volume of distribution (Vd)
Determine whether changes in DNA methylation, histone acetylation, and/or gene expression correlates with clinical response to oral 5-azacitidine and romidepsin | Weekly during cycle 1 and at the start of each subsequent cycle while on study

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Cancer Center @ Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Gaillard SL, Zahurak M, Sharma A, Durham JN, Reiss KA, Sartorius-Mergenthaler S, Downs M, Anders NM, Ahuja N, Rudek MA, Azad N. A phase 1 trial of the oral DNA methyltransferase inhibitor CC-486 and the histone deacetylase inhibitor romidepsin in advanced solid tumors. Cancer. 2019 Aug 15;125(16):2837-2845. doi: 10.1002/cncr.32138. Epub 2019 Apr 23. PMID 31012962